CLINICAL TRIAL: NCT00798343
Title: Evaluation of Heterosubtypic Immune Responses in Older People Before and After Seasonal and Pandemic Influenza Vaccination
Brief Title: Heterosubtypic Immune Responses to Influenza in Older People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Public Health England (Other Government); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UHL10548; MRC 82292
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-06

CONDITIONS: Influenza
Keywords: Influenza, heterosubtypic immune responses
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Seasonal vaccine (Active Comparator): Seasonal influenza vaccination
  Interventions: Biological: Seasonal vaccine
- Pandemic vaccine (Experimental): MF59-adjuvanted H5N1 monovalent vaccine
  Interventions: Biological: H5 vaccine

INTERVENTIONS:
Biological: Seasonal vaccine — Non-adjuvanted seasonal influenza vaccine (total dose 45ug)
  Other Names: Aggripal
  Arms: Seasonal vaccine
Biological: H5 vaccine — MF59-adjuvanted A/Vietnam/1194 H5N1 vaccine 7.5ug dose
  Other Names: Aflunov
  Arms: Pandemic vaccine

SUMMARY:
Vaccination is the principal means of combating epidemic and pandemic influenza. As vaccines induce relatively strain-specific and short-lived antibody responses, annual immunisation with regularly updated vaccine is recommended for seasonal influenza, but would not be expected to protect against a pandemic event. In clinical trials among young adults, at least two doses of avian influenza H5 or H9 subunit vaccine are needed to induce moderate antibody responses. However, studies including older subjects have unexpectedly found that some people aged over 65 yrs have pre-vaccination neutralising antibody to influenza H5 and H9 respectively. These subjects mount a robust antibody response to single dose H5 or H9 pandemic vaccine, suggesting that they are effectively primed to at least some strains of avian influenza.

This exploratory proposal focuses on those elderly subjects whose immune systems already exhibit antibodies to H5 with a goal of investigating the humoral and cellular basis of the immune response to seasonal and pandemic vaccination. We will examine neutralising antibody responses to a range of human and non-human influenza viruses before and after seasonal and pandemic vaccination and evaluate cellular B and T cell immune responses before and after pandemic H5 vaccination

DETAILED DESCRIPTION:
STUDY OBJECTIVES:

Immunological objectives

* To evaluate heterosubtypic neutralising antibody to influenza viruses in older people
* To evaluate heterosubtypic neutralising antibody responses to human and non-human influenza viruses following seasonal influenza vaccine
* To evaluate homologous and heterosubtypic neutralising antibody responses to human and non-human influenza viruses after MF59-adjuvanted H5N1 vaccine;
* To evaluate cellular B and T cell responses to influenza H5 in non-exposed subjects who exhibit anti-H5 neutralising antibodies before and after seasonal (TIV) or pandemic H5 vaccination
* To identify epitopes on the influenza haemagglutinin to which anti-H5 neutralising antibodies in sera from non-exposed subjects are directed Safety Objectives
* To evaluate safety of one or two IM doses of MF59-adjuvanted A/Vietnam/1194/2004 (H5N1) influenza vaccine, containing 7.5 μg of H5 antigen in adult subjects
* To evaluate safety of one IM dose of seasonal influenza vaccine, containing 15 μg of H1, H3 and B antigen in adult subjects

Hypotheses:

* Heterosubtypic cross reacting antibodies to influenza exist in some elderly subjects and can be boosted by a single dose of (a) seasonal TIV or (b) pandemic influenza vaccination
* Heterosubtypic cross reacting antibodies to influenza do not exist in younger subjects and cannot be induced by (a) seasonal TIV or (b) pandemic influenza vaccination

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged over 18 years of age, mentally competent, who have signed an informed consent form after having received a detailed explanation of the study protocol;
2. Subjects willing to be enrolled in the vaccine study if appropriate from prescreening blood test results
3. In good health as determined by:

   1. medical history,
   2. physical examination,
   3. clinical judgment of the Investigator;
4. Able to understand and comply with all study procedures and to complete study diaries, can be contacted, and will be available for study visits

Exclusion Criteria:

1. Receipt of another investigational agent within 4 weeks, or before completion of the safety follow-up period in another study, whichever is longer, prior to enrollment and unwilling to refuse participation in another clinical study through the end of the study;
2. Subjects who experienced any acute disease or infection requiring systemic antibiotic or antiviral therapy (chronic antibiotic therapy for urinary tract prophylaxis is acceptable) within the past 7 days before Visit 1 or any visit where trial vaccination is planned;
3. Subjects who experienced fever (within 3 days prior to Visit 1;
4. Subjects who are pregnant or breastfeeding;
5. Females of childbearing potential who refuse to use an acceptable method of birth control for the duration of the study.
6. Subjects with any serious disease, such as:

   1. cancer,
   2. autoimmune disease (including rheumatoid arthritis),
   3. progressive chronic pulmonary disease (stable controlled respiratory disease including asthma is allowed),
   4. acute or progressive hepatic disease,
   5. acute or progressive renal disease;
7. Subjects for whom elective surgery is planned during the study period;
8. Subjects with bleeding diathesis;
9. Subjects with hypersensitivity to eggs, chicken protein, chicken feathers, influenza viral protein, neomycin or polymyxin or any other component of the study vaccine;
10. Subjects with a history of any neurological symptoms or signs, or anaphylactic shock following administration of any vaccine;
11. Subjects with known or suspected impairment/alteration of immune function, for example, resulting from:

    1. receipt of immunosuppressive therapy (any corticosteroid therapy or cancer chemotherapy),
    2. receipt of immunostimulants,
    3. receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within 3 months prior to Visit 1 or planned during the full length of the study,
    4. high risk for developing an immunocompromising disease;
12. Receipt of another vaccine within 3 weeks prior to Visit 1 or planned vaccination within 3 weeks following the last study vaccination;
13. Subjects with a history of (or current) drug or alcohol abuse that in the investigator's opinion would interfere with safety of the subject or the evaluation of study objectives;
14. Subjects with any condition, which, in the opinion of the Investigator, might interfere with the evaluation of the study objectives.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2009-01; Primary Completion 2010-03 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Neutralising antibody to influenza subtypes | 18 months

SECONDARY OUTCOMES:
Reactogenicity (local and systemic) to H5N1 vaccine | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Iain Stephenson, FRCP, Principal Investigator — University of Leicester
Locations (1):
- University Hospitals Leicester, Leicester, Leicestershire, United Kingdom